CLINICAL TRIAL: NCT06982807
Title: Clinical Study of SMILE 4.0-VISULYZE in Correcting Refractive Errors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-K270
Record Dates: First submitted 2025-05-12; First posted 2025-05-21 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Refractive Surgery; Myopia; Refractive Error
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 4.0-VISULYZE group (Experimental): The 4.0-VISULYZE group had their infusion rates precisely calibrated using 4.0-VISULYZE
  Interventions: Procedure: Group 4.0-VISULYZE
- traditional group (Active Comparator): The traditional group had their infusion rates based on past experience.
  Interventions: Procedure: traditional group

INTERVENTIONS:
Procedure: Group 4.0-VISULYZE — The 4.0-VISULYZE group had their infusion rates precisely calibrated using 4.0-VISULYZE
  Arms: Group 4.0-VISULYZE group
Procedure: traditional group — The traditional group had their infusion rates based on past experience.
  Arms: traditional group

SUMMARY:
The aim of this study is to further optimize the surgical input parameters for patients undergoing Small Incision Lenticule Extraction (SMILE) using the regression model established by the SMILE 4.0-VISULYZE system, thereby achieving satisfactory postoperative refractive outcomes.

In this study, patients scheduled for SMILE surgery at the investigators' hospital will be divided into two groups: a conventional group, where the input parameters are adjusted based on historical experience according to the patient's refractive error, and a 4.0-VISULYZE group, where the input parameters are optimized using the SMILE 4.0-VISULYZE system.

The investigators will compare the postoperative outcomes between the two groups, including uncorrected visual acuity (UCVA), best-corrected visual acuity (BCVA), spherical power, cylindrical power, spherical equivalent (SE), and the proportions of patients achieving postoperative visual acuity ≥0.8, ≥1.0, and ≥1.2 at 1 day, 10 days, 1 month, 3 months, 6 months, and 1 year post-surgery. Additionally, the investigators will evaluate the proportions of patients with postoperative SE within ±0.50D and ±1.0D, as well as postoperative cylindrical power within ±0.50D and ±1.0D, to assess the efficacy and safety of the SMILE 4.0-VISULYZE system in treating refractive errors.

ELIGIBILITY:
Inclusion Criteria:

1. The diopter is relatively stable (the diopter increases within -0.50D per year for 2 consecutive years);
2. Age: 18 to 40 years old;
3. Optimal preoperative corrected visual acuity ≥4.8;
4. More than 2 weeks for soft contact lenses and more than 3 months for hard contact lenses before surgery
5. Patients who are willing to perform SMILE surgery

Exclusion Criteria:

1. Patients with history of eye surgery and trauma;
2. Patients with keratoconus tendency;
3. systemic connective tissue diseases and autoimmune diseases;
4. Patients with high blood pressure, diabetes and heart disease history;
5. Other eye disease history such as uveitis, scleritis and other eye inflammation patients;
6. Patients with scar constitution.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
spherical equivalent | preoperative, postoperative 10 days, 1, 3, 6, 12 months
  Use autorefractor-keratometer and phoroptor to measure degree of myopia and astigmatism，then derive the spherical equivalent.

SECONDARY OUTCOMES:
uncorrected distance visual acuity | preoperative, postoperative 10 days, 1, 3, 6, 12 months
  Use a standardized visual acuity chart (e.g., Snellen or LogMAR chart)
corrected distance visualacuity | preoperative, postoperative 10 days, 1, 3, 6, 12 months
  Use autorefractor-keratometer and phoroptor

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Nantong University, Nantong, Jiangsu, China